CLINICAL TRIAL: NCT04773587
Title: A Phase 3, 4-Week, Parallel Group, Double Blind, Vehicle-Controlled Study of the Safety and Efficacy of ARQ-151 Cream 0.15% Administered QD in Subjects With Atopic Dermatitis
Brief Title: Trial of PDE4 Inhibition With Roflumilast for the Management of Atopic Dermatitis
Acronym: INTEGUMENT-I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARQ-151-311
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Atopic Dermatitis Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Roflumilast Cream 0.15% (Experimental): Participants with mild to moderate AD apply roflumilast cream 0.15% QD for 4 weeks.
  Interventions: Drug: Roflumilast Cream 0.15%
- Vehicle Cream (Placebo Comparator): Participants with mild to moderate AD applied vehicle cream QD for 4 weeks.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Roflumilast Cream 0.15% — Roflumilast Cream 0.15% - Active
  Other Names: ARQ-151
  Arms: Roflumilast Cream 0.15%
Drug: Vehicle Cream — Cream - Vehicle
  Arms: Vehicle Cream

SUMMARY:
This is a parallel group, double blind, vehicle-controlled study to assess the safety and efficacy of roflumilast (ARQ-151) cream vs vehicle applied once daily (qd) for 4 weeks by participants with atopic dermatitis (eczema).

ELIGIBILITY:
Inclusion Criteria:

1. Participants legally competent to sign and give informed consent and, if appropriate, assent as required by local laws.
2. Males and females, ages 6 years and older at time of signing Informed Consent (Screening). Only subjects 18 years and older will be enrolled at sites located in the province of Québec in Canada.
3. Diagnosed with atopic dermatitis 6 months duration (3 months for children), as determined by the Investigator. Stable disease for the past 4 weeks with no significant flares in atopic dermatitis before screening.
4. Females of childbearing potential (FOCBP) must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline/Day 1. In addition, sexually active FOCBP must agree to use at least one form of a highly effective or barrier method of contraception throughout the trial.
5. In good health as judged by the Investigator.
6. Subjects considered reliable and capable of adhering to the Protocol and visit schedule, according to the judgment of the Investigator.

Exclusion Criteria:

1. Subjects with any serious medical condition or clinically significant abnormality that would prevent study participation or place the subject at significant risk, as judged by the Investigator
2. Has unstable AD or any consistent requirement for high potency topical steroids.
3. Subjects who are unwilling to refrain from prolonged sun exposure and from using a tanning bed or other artificial light emitting devices (LEDs) for 4 weeks prior to Baseline/Day 1 and during the study.
4. Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.
5. Previous treatment with ARQ-151.
6. Subjects with a history of chronic alcohol or drug abuse within 6 months prior to Screening.
7. Parent(s)/legal guardian(s) who are unable to communicate, read, or understand the local language(s). Subjects who are unable to communicate, read or understand the local language, or who display another condition, which in the Investigator's opinion, makes them unsuitable for clinical study participation.
8. Subjects who are family members of the clinical study site, clinical study staff, or sponsor, or family members of enrolled subjects living in the same house.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (49):
- United States (42):
  - Arcutis Clinical Site 57, Montgomery, Alabama
  - Arcutis Clinical Site 34, Scottsdale, Arizona
  - Arcutis Clinical Site 58, Little Rock, Arkansas
  - Arcutis Clinical Site 40, Beverly Hills, California
  - Arcutis Clinical Site 06, Encinitas, California
  - Arcutis Clinical Site 52, Los Angeles, California
  - Arcutis Clinical Site 05, San Diego, California
  - Arcutis Clinical Site 08, San Francisco, California
  - Arcutis Clinical Site 62, Thousand Oaks, California
  - Arcutis Clinical Site 30, Coral Gables, Florida
  - Arcutis Clinical Site 04, Jacksonville, Florida
  - Arcutis Clinical Site 15, Largo, Florida
  - Arcutis Clinical Site 39, Miami Lakes, Florida
  - Arcutis Clinical Site 38, North Miami Beach, Florida
  - Arcutis Clinical Site 01, Tampa, Florida
  - Arcutis Clinical Site 61, Wellington, Florida
  - Arcutis Clinical Site 26, Sandy Springs, Georgia
  - Arcutis Clinical Site 13, Rolling Meadows, Illinois
  - Arcutis Clinical Site 48, Clarksville, Indiana
  - Arcutis Clinical Site 02, Indianapolis, Indiana
  - Arcutis Clinical Site 03, Louisville, Kentucky
  - Arcutis Clinical Site 36, Rockville, Maryland
  - Arcutis Clinical Site 55, Auburn Hills, Michigan
  - Arcutis Clinical Site 54, Bay City, Michigan
  - Arcutis Clinical Site 46, Clarkston, Michigan
  - Arcutis Clinical Site 37, Detroit, Michigan
  - Arcutis Clinical Site 10, New Brighton, Minnesota
  - Arcutis Clinical Site 33, Reno, Nevada
  - Arcutis Clinical Site 42, East Windsor, New Jersey
  - Arcutis Clinical Site 17, Gresham, Oregon
  - Arcutis Clinical Site 16, Portland, Oregon
  - Arcutis Clinical Site 14, Portland, Oregon
  - Arcutis Clinical Site 35, Newtown Square, Pennsylvania
  - Arcutis Clinical Site 101, Johnston, Rhode Island
  - Arcutis Clinical Site 31, Murfreesboro, Tennessee
  - Arcutis Clinical Site 19, Arlington, Texas
  - Arcutis Clinical Site 43, Bellaire, Texas
  - Arcutis Clinical Site 27, Houston, Texas
  - Arcutis Clinical Site 20, Houston, Texas
  - Arcutis Clinical Site 28, San Antonio, Texas
  - Arcutis Clinical Site 21, South Jordan, Utah
  - Arcutis Clinical Site 12, Spokane, Washington
- Canada (7):
  - Arcutis Clinical Site 41, Calgary, Alberta
  - Arcutis Clinical Site 29, Fredericton, New Brunswick
  - Arcutis Clinical Site 11, Markham, Ontario
  - Clinical Site 25, Mississauga, Ontario
  - Arcutis Clinical Site 32, Peterborough, Ontario
  - Arcutis Clinical Site 09, Windsor, Ontario
  - Arcutis Clinical Site 24, Montreal, Quebec

REFERENCES:
- [Derived] Simpson EL, Eichenfield LF, Alonso-Llamazares J, Draelos ZD, Ferris LK, Forman SB, Gooderham M, Gonzalez ME, Hebert AA, Kircik LH, Lomaga M, Moore A, Papp KA, Prajapati VH, Hanna D, Snyder S, Krupa D, Burnett P, Almaraz E, Higham RC, Chu DH, Berk DR. Roflumilast Cream, 0.15%, for Atopic Dermatitis in Adults and Children: INTEGUMENT-1 and INTEGUMENT-2 Randomized Clinical Trials. JAMA Dermatol. 2024 Nov 1;160(11):1161-1170. doi: 10.1001/jamadermatol.2024.3121. PMID 39292443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 65 centers in the United States, Canada, and Poland.
Groups:
- Roflumilast Cream 0.15%: Participants with mild to moderate AD applied roflumilast cream 0.15% once daily (QD) for 4 weeks.
Period: Overall Study
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Started | 433 | 221
Completed | 404 | 208
Not Completed | 29 | 13
Not completed — Lost to Follow-up | 11 | 3
Not completed — Adverse Event | 6 | 3
Not completed — Lack of Efficacy | 5 | 2
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Noncompliance | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Consent withdrawn due to AEs of nausea, headaches, dizziness, and brain fog | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream | Total
Number analyzed (Participants) | 433 | 221 | 654
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (19.14) | 28.5 (18.94) | 28.2 (19.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 237 | 129 | 366
  Male | 196 | 92 | 288
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 99 | 56 | 155
  Not Hispanic or Latino | 333 | 164 | 497
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 261 | 129 | 390
  American Indian or Alaska native | 2 | 0 | 2
  Asian | 63 | 32 | 95
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  Black or African American | 80 | 46 | 126
  Multiple | 12 | 6 | 18
  Other | 14 | 8 | 22
Randomization validated Investigator's Global Assessment Scale for Atopic Dermatitis (vIGA-AD) [Count of Participants; unit: Participants] — The vIGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (reported only in integers of 0 to 4 where 0 is clear), with higher scores indicative of greater symptom severity.
  Participants
    2 - Mild | 105 | 57 | 162
    3 - Moderate | 328 | 164 | 492
Verified vIGA-AD [Count of Participants; unit: Participants] — The vIGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (reported only in integers of 0 to 4 where 0 is clear), with higher scores indicative of greater symptom severity.
  Participants
    Mild | 103 | 59 | 162
    Moderate | 330 | 162 | 492

OUTCOME MEASURES:

1. Primary Outcome: Achievement of Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) Success at Week 4
Description: The percentage of participants achieving vIGA-AD "success" is presented with multiple imputation of missing observations. vIGA-AD "success" is defined as a vIGA-AD score of 'clear' or 'almost clear' PLUS a 2-grade improvement from Baseline. The vIGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (reported only in integers of 0 to 4 where 0 is clear), with higher scores indicative of greater symptom severity.
Time Frame: Week 4
Population: All randomized participants are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 433 | 221
percentage of participants | 32.0 [27.79 to 36.63] | 15.2 [11.06 to 20.64]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference in vIGA-AD Success at Week 4; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations; Odds Ratio (OR) = 2.96, 95% CI 2-sided [1.881 to 4.647] — Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations

2. Secondary Outcome: Achievement of vIGA-AD Success at Week 4 in Participants With "Moderate" Baseline Scores
Description: The percentage of participants with moderate baseline scores achieving vIGA-AD "success" is presented with multiple imputation of missing observations. vIGA-AD "success" is defined as a vIGA-AD score of 'clear' or 'almost clear' PLUS a 2-grade improvement from Baseline in participants with a 'moderate' baseline vIGA-AD score. The vIGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (0 'clear' to 4 'severe'), with higher scores indicative of greater symptom severity.
Time Frame: Week 4
Population: All randomized participants who were included in the "moderate" baseline vIGA-AD group during randomization are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Roflumilast Cream 0.15%: Participants with moderate AD applied roflumilast cream 0.15% once daily (QD) for 4 weeks.
- Vehicle Cream: Participants with moderate AD applied vehicle cream QD for 4 weeks.
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 328 | 164
percentage of participants | 35.0 [29.97 to 40.36] | 17.5 [12.38 to 24.13]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference in vIGA-AD Success at Week 4; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site with multiple imputation of missing observations; Odds Ratio (OR) = 2.67, 95% CI 2-sided [1.640 to 4.359] — Stratified by pooled study site with multiple imputation of missing observations

3. Secondary Outcome: Achievement of a 4-Point Reduction in the Average, Weekly Worst Itch Numeric Rating Scale (WI-NRS) at Week 4 in Participants ≥12 Years of Age With Baseline WI-NRS ≥ 4
Description: The percentage of participants ≥12 years of age with a baseline WI-NRS ≥4 achieving WI-NRS success at Week 4 is presented with multiple imputation of missing observations. The WI-NRS is a simple, single item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the participant experienced in the previous 24 hours (higher scores indicate higher itch severity).
Time Frame: Week 4
Population: All randomized participants ≥12 years of age with a baseline WI-NRS ≥4 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 278 | 135
percentage of participants | 33.6 [28.19 to 39.41] | 20.7 [14.61 to 28.58]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; WI-NRS Success at Week 4; Test type: Superiority; p = 0.0089, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations; Odds Ratio (OR) = 1.98, 95% CI 2-sided [1.186 to 3.319] — Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations

4. Secondary Outcome: Achievement of a 4-Point Reduction in the Average, Weekly WI-NRS at Week 2 in Participants ≥12 Years of Age With Baseline WI-NRS ≥ 4
Description: The percentage of participants ≥12 years of age with a baseline WI-NRS ≥4 achieving WI-NRS success at Week 2 is presented with multiple imputation of missing observations. The WI-NRS is a simple, single item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the participant experienced in the previous 24 hours (higher scores indicate higher itch severity).
Time Frame: Week 2
Population: All randomized participants ≥12 years of age with a baseline WI-NRS ≥4 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 278 | 135
percentage of participants | 23.8 [19.14 to 29.24] | 9.8 [5.79 to 16.03]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15%; WI-NRS Success at Week 2; Test type: Superiority; p = 0.0016, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations; Odds Ratio (OR) = 2.81, 95% CI 2-sided [1.450 to 5.457] — Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations

5. Secondary Outcome: Achievement of a 4-Point Reduction in the Average, Weekly WI-NRS at Week 1 in Participants ≥12 Years of Age With Baseline WI-NRS ≥ 4
Description: The percentage of participants ≥12 years of age with a baseline WI-NRS ≥4 achieving WI-NRS success at Week 1 is presented with multiple imputation of missing observations. The WI-NRS is a simple, single item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the participant experienced in the previous 24 hours (higher scores indicate higher itch severity).
Time Frame: Week 1
Population: All randomized participants ≥12 years of age with a baseline WI-NRS ≥4 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 278 | 135
percentage of participants | 9.5 [6.60 to 13.60] | 2.3 [0.77 to 6.41]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; WI-NRS Success at Week 1; Test type: Superiority; p = 0.0159, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations; Odds Ratio (OR) = 3.81, 95% CI 2-sided [1.161 to 12.511] — Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations

6. Secondary Outcome: Achievement of ≥ 75% Reduction in the Eczema Area and Severity Index (EASI-75) at Week 4
Description: The percentage of participants achieving EASI-75 is presented with multiple imputation of missing observations. EASI-75 is a ≥75% reduction from the baseline EASI score. EASI combines the assessment of the severity of lesions and the area affected into a single total score in the range 0 (no disease) to 72 (maximal disease). To calculate the EASI, the sum of the severity rating (0 to 3 with 3 being the most severe) for four clinical signs are multiplied with the numerical value of the area affected and with the percentage of the four body areas.
Time Frame: Week 4
Population: All randomized participants are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 433 | 221
percentage of participants | 43.2 [38.54 to 47.94] | 22.0 [16.97 to 28.04]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; EASI-75 at Week 4; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations; Odds Ratio (OR) = 3.17, 95% CI 2-sided [2.102 to 4.795] — Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations

7. Secondary Outcome: Achievement of vIGA-AD Score of 'Clear' or 'Almost Clear' at Week 4
Description: The percentage of participants scoring 'clear' or 'almost clear' on vIGA-AD at Week 4 is presented with multiple imputation of missing observations. The vIGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (0 'clear' to 4 'severe'), with higher scores indicative of greater symptom severity.
Time Frame: Week 4
Population: All randomized participants are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 433 | 221
percentage of participants | 41.5 [36.93 to 46.25] | 25.2 [19.91 to 31.41]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; vIGA-AD Score of 'Clear' or 'Almost Clear' at Week 4; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations; Odds Ratio (OR) = 2.56, 95% CI 2-sided [1.707 to 3.843] — Stratified by pooled study stie and vIGA-AD randomization strata with multiple imputation of missing observations

8. Secondary Outcome: Achievement of vIGA-AD Success at Week 2
Description: The percentage of participants achieving "success" on the VIGA-AD at Week 2 is presented with multiple imputation of missing observations. vIGA-AD "success" is defined as a vIGA-AD score of 'clear' or 'almost clear' PLUS a 2-grade improvement from Baseline. The vIGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (0 'clear' to 4 'severe'), with higher scores indicative of greater symptom severity.
Time Frame: Week 2
Population: All randomized participants are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 433 | 221
percentage of participants | 21.2 [17.57 to 25.33] | 6.4 [3.84 to 10.44]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; vIGA-AD Success at Week 2; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations; Odds Ratio (OR) = 4.28, 95% CI 2-sided [2.310 to 7.926] — Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations

9. Secondary Outcome: Achievement of vIGA-AD Success at Week 1
Description: The percentage of participants achieving "success" on the VIGA-AD at Week 1 is presented with multiple imputation of missing observations. vIGA-AD "success" is defined as a vIGA-AD score of 'clear' or 'almost clear' PLUS a 2-grade improvement from Baseline. The vIGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (0 'clear' to 4 'severe'), with higher scores indicative of greater symptom severity.
Time Frame: Week 1
Population: All randomized participants are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 433 | 221
percentage of participants | 8.1 [5.87 to 11.03] | 0.5 [0.08 to 2.52]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; vIGA-AD Success at Week 1; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations; Odds Ratio (OR) = 25.41, 95% CI 2-sided [2.815 to 229.388] — Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations

10. Secondary Outcome: Achievement of vIGA-AD Score of 'Clear' or 'Almost Clear' at Week 2
Description: as for outcome 7
Time Frame: Week 2
Population: All randomized participants are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 433 | 221
percentage of participants | 31.8 [27.58 to 36.38] | 13.6 [9.72 to 18.79]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; vIGA-AD Score of 'Clear' or 'Almost Clear' at Week 2; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations; Odds Ratio (OR) = 3.62, 95% CI 2-sided [2.217 to 5.911] — Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations

11. Secondary Outcome: Achievement of vIGA-AD Score of 'Clear' or 'Almost Clear' at Week 1
Description: as for outcome 7
Time Frame: Week 1
Population: All randomized participants are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 433 | 221
percentage of participants | 14.3 [11.33 to 17.93] | 5.9 [3.47 to 9.80]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; vIGA-AD Score of 'Clear' or 'Almost Clear' at Week 1; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations; Odds Ratio (OR) = 3.46, 95% CI 2-sided [1.705 to 7.007] — Stratified by pooled study site and vIGA-AD randomization strata with multiple imputation of missing observations

ADVERSE EVENTS:
Time Frame: Up to approximately 29 days
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/433 | 0/221
Serious Adverse Events (participants affected / at risk) | 4/433 | 0/221
Other Adverse Events (participants affected / at risk) | 0/433 | 0/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast Cream 0.15% (N=433) | Vehicle Cream (N=221)
Diverticulitis (Infections and infestations) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Pulmonary embolism (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor is generally supportive of publication of trial results.

DOCUMENTS (2):
  • Study Protocol (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT04773587/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT04773587/SAP_002.pdf